CLINICAL TRIAL: NCT05316896
Title: Investigation of the Efficacy of Internal and External Perturbation Exercises on Functional Parameters in Stroke Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Nagihan Bodur, Physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MedipolUni
Record Dates: First submitted 2022-03-08; First posted 2022-04-07 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal perturbation (Experimental): The people included in this group did 6 internal perturbation exercises with 10 repetitions in each session. The patients performed a total of 60 perturbation exercises in one session. Perturbations were chosen according to the patient's tolerance, from easy to difficult. Treatment protocols of stroke individuals were determined according to their functional levels. 6 of the exercises given below were chosen according to the levels determined at the beginning of the study and were progressed by getting more difficult.
  Interventions: Other: Internal Perturbation
- Eksternal perturbation (Experimental): The individuals included in this group performed 6 external perturbation exercises with 10 repetitions in each session. The patients performed a total of 60 perturbation exercises in one session. Perturbations were chosen according to the patient's tolerance, from easy to difficult. Treatment protocols of stroke individuals were determined according to their functional levels. 6 of the exercises given below were chosen according to the levels determined at the beginning of the study and were progressed by getting more difficult.
  Interventions: Other: Eksternal Perturbation

INTERVENTIONS:
Other: Internal Perturbation — * Raising and lowering arms 90 degrees forward and sideways with eyes open and closed.
  * In tandem stance with eyes open and closed, arms are raised and lowered 90 degrees forward and to the side.
  * While standing on one leg with eyes open and closed, arms are raised and lowered 90 degrees forward and to the side.
  * Step forward and backward with right and left foot alternately
  * Take a step back and step back alternately with right and left foot
  * Put the right foot on the step and take it back, then do the same with the left foot and ask the patient to do it quickly.
  * First step on the step with the right foot and put the left foot next to it, then step down with the right foot and take the left foot with it, repeat the same with the left foot and ask the patient to do this. rapidly.
  * Normal gait, sideways gait, tandem gait, backward gait, raising and lowering the arms forward and sideways 90 degrees, respectively, during back-to-back tandem gait.
  Arms: Internal perturbation
Other: Eksternal Perturbation — * Front, side, and rear loading and release, pushing and pulling while standing with eyes open and closed
  * Front, side and rear loading and release, pushing and pulling while standing in tandem with eyes open and closed
  * Loading and releasing from the front, sides and back, pushing and pulling while turning the head left and right while standing
  * Front, side and rear loading and release, pushing and pulling while standing up and down with eyes open and closed
  * Front, side, and rear loading and release, pushing and pulling while standing on one leg with eyes open and closed
  * Holding the ball thrown by physiotherapist
  * Kicking a ball thrown by physiotherapist
  * Holding the ball thrown by the physiotherapist while standing in tandem, walking, walking sideways, walking in tandem, walking backwards.
  Arms: Eksternal perturbation

SUMMARY:
Stroke is a serious medical condition that causes the death of brain cells as a result of blockage of a blood vessel that feeds the brain (ischemic stroke) or bleeding in or around the brain (hemorrhagic stroke). People who have had a stroke have a higher risk of falling than people who have not had a stroke at the same age. Lack of balance control not only increases the risk of falling, but also leads to fear of falling and reduces the integration of people with stroke into society.

The central nervous system uses two main postural strategies to maintain and restore balance when perturbed. These; are anticipatory and compensatory postural adjustments. Anticipatory postural adjustments control the position of the body's center of mass by activating the trunk and leg muscles prior to a forthcoming body perturbation, thus minimizing the risk of loosing equilibrium. Compensatory postural adjustment are initiated by sensory feedback signals and serve as a mechanism of restoration of the position of the center of mass after a perturbation has already occurred.

In this study, the investigators aimed to determine which one is more effective, unlike previous studies that showed that internal and external perturbation exercises were effective when applied together. For this purpose, the researchers the planned to investigate and compare the effects on balance, performance, activity and participation in individuals to whom only internal perturbations were applied and only external perturbations were applied.

The participants will be divided into 2 groups, as Group A and Group B, with 10 participants in each group, in a randomized controlled manner.

Treatment Protocol:

Conventional treatment was applied to participants included in both groups for 4 weeks, 5 days a week, 40-minute sessions. In addition to conventional treatment, 30 minutes of perturbation-based balance training was given to the participant in the study. Participants in Group A received internal perturbation training, and participants in Group B received external perturbation training.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral stroke history
* Adults with chronic stroke (>6 months poststroke)
* Ability to stand for at least 30 seconds without support

Exclusion Criteria:

* Those with Parkinson's disease, amputation, severe osteoporosis
* Those with uncontrolled diabetes, hypertension
* In addition to stroke, the presence of any problem that may adversely affect balance
* Areas below 24 in the mini mental state test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-11-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in dynamic and static balance on the Berg Balance Scale at 4 weeks | baseline and 4 weeks
  Berg balance scale is a valid and reliable test that measures both dynamic and static balance. It evaluates the body's ability to maintain position during 14 different activities in which the support surface decreases and the center of gravity changes, by observation. It is scored between 0-4 points, while at 0 the activity cannot be completed, at 4 it is completed independently. The total score is 56. If the score obtained at the end of the test is between 0-20, it is interpreted as poor balance skills, between 21-40 as acceptable balance and between 41-56 as advanced balance skills.
Change from baseline in balance on the Timed Up and Go Test at 4 weeks | baseline and 4 weeks
  For the timed up and go test, the patient gets up from the chair without arm support, walks 3 meters, returns and sits back in the chair. The total time it takes to complete the test is recorded in seconds using a stopwatch. The evaluation results are valid as they include maneuvers used in daily life. Individuals with independent balance and mobility skills complete the test in less than 10 seconds, individuals who complete it in more than 30 seconds are dependent on many activities and mobility skills in daily life.
Change from baseline in balance 10-meter Walking Test at 4 weeks | baseline and 4 weeks
  In this test, the person is asked to walk at his own normal pace in a pre-measured 10-meter area. The time starts when the person's foot is on the starting line and ends when they cross the finish line. Two measurements are made and the best value is recorded in meters/second.
Change from baseline in balance on the One Leg Standing Test at 4 weeks | baseline and 4 weeks
  One foot is lifted so that it does not touch the other leg and the time is measured with a stopwatch. At first the eyes are open. When the eye open test is completed, the test is done with the eyes closed and it is expected that he can maintain his balance for 30 seconds. An imbalance is considered if the lifted leg touches the other leg, the foot touches the floor, bounces or bounces, or anything in the environment is touched for support.

SECONDARY OUTCOMES:
Change from baseline in daily life activities on the Nottingham Health Profile at 4 weeks | baseline and 4 weeks
  It is a measurement tool that evaluates the health problems of individuals and how these problems affect their daily activities. Scale; It consists of 6 parameters and 38 items in total. Parameters; energy (3 items), pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items), and physical activity (8 items). The answers are yes-no. The score weight of each question is different. Each field is scored between 0-100. The higher the score, the worse the health condition.
Change from baseline in ambulation ability on the Functional Ambulation Classification (FAS) at 4 weeks | baseline and 4 weeks
  It is a scale that evaluates the ambulation ability of patients. It is divided into six categories, graded from 0 to 5: FAS 0: no ambulation, FAS 1-2: a person cannot walk without support, FAS 3-5: able to walk 6 meters on their own.
Motor development in stroke patients on the Brunnstrom Hemiplegia Recovery Staging at baseline | baseline
  It is a short and easily applicable staging system for evaluating motor development in stroke patients. Motor development is defined as 6 stages. The lowest, flaccid period without voluntary movements is considered stage 1, and the presence of isolated movements is considered stage 6. Upper, lower extremity and hand are evaluated separately
Assessment method for spasticity on the Modified Ashworth Scale at baseline | baseline
  It is the most commonly used assessment method for spasticity in the international platform. The patient is examined in a supine and relaxed position. The joint is moved passively, repetitively and rapidly, and the resistance is staged between 0-4 according to the examination findings.0; no increase in tone 1; there is a slight increase in muscle tone, minimal resistance is felt at the end of the movement when the affected part is flexed or extended 1+; resistance during movement is felt in less than half of joint movement 2; resistance is felt during most joint movement, but the affected part is easily moved 3; passive movement throughout the range of motion is difficult 4; the affected part is rigid in flexion or extension.
Change from baseline in level of disability on the Barthel Index at 4 weeks | baseline and 4 weeks
  It is used to measure the level of disability experienced by the patient during activities of daily living. It consists of a total of 10 main items. Nutrition, wheelchair-bed transfer, self-care, sitting on the toilet, washing, walking on a smooth surface, going up and down stairs, dressing, undressing, bowel and bladder care are questioned. The total score is evaluated between 0 and 100. 0-20 points: fully dependent, 21-61 points: severely dependent, 62-90 points: moderately dependent, 91-99: mildly dependent, 100 points: fully independent.
Change from baseline in quality of life on the Stroke Impact Scale at 4 weeks | baseline and 4 weeks
  It is a stroke-specific health-related quality of life scale. There are 59 items in 8 areas. 4 items on strength, 5 items on hand function, 9 items on mobility, 10 items on activities of daily living, 7 items on memory, 9 items on mood, 7 items on communication, and 8 items on social participation. contains substance. The score for each section ranges from 0-100. A high score means a high quality of life. In addition to 8 subsections, it includes the evaluation of the perception of recovery after stroke with a 0-100 point visual analog scale (0: no recovery, 100: complete recovery).
Change from baseline in balance on the 4-Step Climbing Test at 4 weeks | baseline and 4 weeks
  Participants are instructed to go up and down a 4-step ladder as quickly as possible. The time to go up and down 4 digits is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University Sefakoy Hospital, Istanbul, Turkey (Türkiye)